CLINICAL TRIAL: NCT03482388
Title: A Crowdsourced Intervention to Promote Hepatitis B and C Testing Among Men Who Have Sex With Men in China: a Nationwide Online Randomized Controlled Trial
Brief Title: Crowdsourcing to Promote HBV and HCV Testing in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Doris Duke Charitable Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 18-0251
Record Dates: First submitted 2018-03-22; First posted 2018-03-29 (Actual); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis; Hepatitis B; Hepatitis C
Keywords: Hepatitis; Hepatitis B; Hepatitis C; Men who have sex with men; Crowdsourcing; China; Testing
MeSH Terms: conditions — Hepatitis; Hepatitis B; Hepatitis C; Homosexuality

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned in a 1:1 ratio to the study intervention or control
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crowdsourced intervention (Experimental): A multimedia component will deliver two videos and two images promoting HBV and HCV testing developed through a crowdsourcing contest in China. A participatory component will invite men to submit suggestions for how to improve crowdsourced videos and images.
  Interventions: Behavioral: Crowdsourced materials
- Control (Other): No images or videos will be viewed, and suggestions for improving hepatitis testing materials will not be collected.
  Interventions: Other: Control

INTERVENTIONS:
Behavioral: Crowdsourced materials — Among participants randomized to the intervention arm, intervention images and videos promoting HBV and HCV testing will be delivered through the WeChat platform. Men will also be invited to submit suggestions for how to improve intervention videos and images.
  Arms: Crowdsourced intervention
Other: Control — Participants will not view any images or videos promoting HBV and HCV testing.
  Arms: Control

SUMMARY:
This is an online randomized controlled trial (RCT) comparing men who have sex with men (MSM) exposed to a crowdsourced intervention to MSM who did not receive the intervention to determine the effect on Hepatitis B Virus (HBV) and Hepatitis C Virus (HCV) testing. Participants will be randomly assigned in a 1:1 ratio to intervention or control using a computer-based allocation system. Participants will be assessed for primary and secondary outcomes four weeks after randomization.

DETAILED DESCRIPTION:
700 MSM will be recruited through social media operated by gay organizations in China. Eligible participants will be born biologically male, age 16 years or older, report previous anal sex with another man, and reside in China. Men self-reporting previous HBV vaccination, HBV testing, or HCV testing will be excluded. After completing a baseline online survey, participants will be randomly assigned to intervention or control arms with a 1:1 allocation ratio. The intervention will include two components: (1) a multimedia component will deliver two videos and two images promoting HBV and HCV testing developed through a crowdsourcing contest in China. (2) A participatory component will invite men to submit suggestions for how to improve crowdsourced videos and images. The control arm will not view any images or videos and will not be invited to submit suggestions. All participants will be offered reimbursement for HBV and HCV testing costs. The primary outcome is HBV and HCV test uptake confirmed through electronic submission of test report photos within four weeks of enrollment. Secondary outcomes include self-reported HBV and HCV test uptake, HBV vaccination uptake, and change in stigma toward people living with HBV measured through a follow-up survey after four weeks. Men with primary and secondary outcomes will be calculated using intention to treat and as-exposed analyses and compared using two-sided 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* 16 years of age or older
* male
* report having had anal sex with another man at least once in the past
* currently reside in China
* willing to provide working mobile phone number and WeChat account

Exclusion Criteria:

* previous HBV vaccination
* previous HBV testing
* previous HCV testing

Min Age: 16 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 700 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2018-06-09 (Actual)

PRIMARY OUTCOMES:
Confirmed HBV and HCV test uptake | enrollment - 4 weeks after enrollment
  Defined as frequency of men who had both HBsAg test uptake and anti-HCV IgG test uptake confirmed through electronic submission of a test report photo showing serology results, age of tester, sex of tester, and date of test

SECONDARY OUTCOMES:
Confirmed HBV test uptake | enrollment - 4 weeks after enrollment
  Defined as frequency of men who had HBsAg test uptake through electronic submission of a test report photo showing serology results, age of tester, sex of tester, and date of test
Confirmed HCV test uptake | enrollment - 4 weeks after enrollment
  Defined as frequency of men who had anti-HCV IgG test uptake confirmed through electronic submission of a test report photo showing serology results, age of tester, sex of tester, and date of test
Self-reported HBV test uptake | enrollment - 4 weeks after enrollment
  Defined as frequency of men who had HBsAg uptake within four weeks of enrollment, self-reported in follow-up survey
Self-reported HCV test uptake | enrollment - 4 weeks after enrollment
  Defined as frequency of men who had anti-HCV IgG uptake within four weeks of enrollment, self-reported in follow-up survey
HBV vaccination uptake | enrollment - 4 weeks after enrollment
  Defined as frequency of men who had receipt of at least a one dose of the HBV vaccine within four weeks of enrollment, self-reported in follow-up survey
HBV vaccination uptake among men with confirmed susceptibility to HBV infection | enrollment - 4 weeks after enrollment
  Defined as frequency of men with negative HBsAg and negative anti-HBs results confirmed through electronic submission of a test report photo showing serology results, who had receipt of at least a one dose of the HBV vaccine within four weeks of enrollment, self-reported in follow-up survey
HIV test uptake | enrollment - 4 weeks after enrollment
  Defined as frequency of men who had HIV test uptake within four weeks of enrollment, self-reported in follow-up survey
Chlamydia test uptake | baseline - 4 weeks after enrollment
  Defined as frequency of men who had chlamydia test uptake within four weeks of enrollment, self-reported in follow-up survey
Gonorrhea test uptake | enrollment - 4 weeks after enrollment
  Defined as frequency of men who had gonorrhea test uptake within four weeks of enrollment, self-reported in follow-up survey
Syphilis test uptake | enrollment - 4 weeks after enrollment
  Defined as frequency of men who had syphilis test uptake within four weeks of enrollment, self-reported in follow-up survey
Change in stigma toward people living with HBV | enrollment - 4 weeks after enrollment
  Continuous variable, defined as difference between Toronto Chinese HBV Stigma Scale score assessed at follow-up and baseline. Stigma toward people living with HBV will be measured at baseline and follow-up using 20 survey items that are each on a five point Likert scale. The 20 items were originally developed as the Toronto Chinese HBV Stigma Scale (potential range of 20 - 100), which has been previously validated and correlated to HBV testing behaviors among Chinese populations. Decreased stigma toward people living with HBV will be defined as a mean composite score that is less at follow-up compared to baseline.
Visit with a physician after hepatitis test uptake | enrollment - 4 weeks after enrollment
  Defined as frequency of men who had HBV and/or HCV test uptake and saw a physician to discuss hepatitis test results within four weeks of enrollment, self-reported in follow-up survey

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Tucker, MD, PhD, MA, Study Director — University of North Carolina, Chapel Hill; Thomas Fitzpatrick, Principal Investigator — Institute for Global Health and Infectious Diseases
Locations (1):
- UNC Project-China, Guangzhou, China

IPD SHARING:
Plan to Share IPD: Yes
All de-identified data generated or analyzed during this study will be included in published articles and supplementary information files.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: They will be shared upon publication of the main manuscript.

REFERENCES:
- [Derived] Palmer MJ, Henschke N, Villanueva G, Maayan N, Bergman H, Glenton C, Lewin S, Fonhus MS, Tamrat T, Mehl GL, Free C. Targeted client communication via mobile devices for improving sexual and reproductive health. Cochrane Database Syst Rev. 2020 Jul 14;8(8):CD013680. doi: 10.1002/14651858.CD013680. PMID 32779730
- [Derived] Fitzpatrick T, Zhou K, Cheng Y, Chan PL, Cui F, Tang W, Mollan KR, Guo W, Tucker JD. A crowdsourced intervention to promote hepatitis B and C testing among men who have sex with men in China: study protocol for a nationwide online randomized controlled trial. BMC Infect Dis. 2018 Sep 29;18(1):489. doi: 10.1186/s12879-018-3403-3. PMID 30268114